CLINICAL TRIAL: NCT02132962
Title: Sarcopenia and Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-4-2012-162
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Biopsy

ARMS (2):
- Healthy controls (Active Comparator): Amino acid infusion
  Interventions: Dietary Supplement: Amino acid infusion; Other: Bloodsamples, Biopsies.
- Cirrhosis (Active Comparator): Amino acid infusion
  Interventions: Dietary Supplement: Amino acid infusion; Other: Bloodsamples, Biopsies.

INTERVENTIONS:
Dietary Supplement: Amino acid infusion
Other: Bloodsamples, Biopsies.

SUMMARY:
The study investigates the effect of aminoacid infusion on proteinturnover in muscle from cirrhosis subjects, compared to healthy controls.

The hypothesis is that aminoacid infusion can attenuate the increase in proteindegradation that follows cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Diagnosis of cirrhosis, Child-Pugh A, B, C.

Exclusion Criteria:

* Acute illness within 3 weeks
* Ascites collections within 10 days
* Heart-, kidney, pulmonary disease. Cancer. Type 1 diabetes.
* Active alkoholdrinking

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Turnover of phenylalanine and tyrosine in skeletal muscle tissue during amino acid infusion. Inflammatory markers. Protein signaling cascade. | 24 weeks
  Using stable isotope tracer technique with infusion of phenylalanine and tyrosine tracer.
  Using ELISA technique. Using PCR and western blot technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark